CLINICAL TRIAL: NCT06587477
Title: Effect of Cancer Treatment on Testicular Function and Semen Quality in Male Childhood and Adolescent Cancer Survivors
Brief Title: Testicular Function and Semen Quality in Male Childhood and Adolescent Cancer Survivors
Status: Recruiting | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other); Hong Kong Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: UW21-038
Record Dates: First submitted 2024-05-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Cancer, Treatment-Related; Late Effect; Semen Analysis
Keywords: cancer treatment; testicular function; semen quality; cancer survivors
MeSH Terms: conditions — Neoplasms, Second Primary | interventions — Semen Analysis; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Biospecimen Retention: Samples Without DNA — Excess serum for future research use
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Male childhood and adolescent cancer survivors: Male childhood and adolescent cancer survivors
  Interventions: Other: Hormonal profile; Other: Semen analysis; Other: Questionnaire
- Controls: Aged-matched controls from men attending the Family Planning Association for premarital check-up
  Interventions: Other: Hormonal profile; Other: Semen analysis; Other: Questionnaire

INTERVENTIONS:
Other: Hormonal profile — Blood for FSH, LH, testosterone
Other: Semen analysis — Semen analysis
Other: Questionnaire — The European Male Ageing Study (EMAS) questionnaire

SUMMARY:
Cancer treatment can affect the testicular function, including sperm and hormonal functions. The aim of this study is to assess the testicular function and semen quality in young men who recover from childhood and adolescent cancer in Hong Kong. This can provide more information for pre-treatment counselling as well as improve post treatment survivorship care. The testicular function will be compared to aged-matched controls from men attending the Family Planning Association for premarital check-up.

DETAILED DESCRIPTION:
This is a cohort observational study. The target population for the trial will be men who have received chemotherapy and/ or radiotherapy for cancer diagnosed when they were < 18 years old, currently > 18 years old to 50 years old and cancer in remission for at least 2 years. The testicular function, including sperm and hormonal functions, will be compared with aged-matched controls from men attending the Family Planning Association for premarital check-up.

ELIGIBILITY:
Inclusion Criteria:

* Men who have received chemotherapy and/ or radiotherapy for cancer diagnosed when they were < 18 years old.
* > 18 years old to 50 years old
* Cancer in remission for at least 2 years

Exclusion Criteria:

* Unable to ejaculate by masturbation to provide semen samples
* Cryptorchidism, testicular cancer, history of vasectomy
* On testosterone replacement therapy
* Refusal to join the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Target participant Population
  * The target population for the trial will be men who have received chemotherapy and/ or radiotherapy for cancer diagnosed when they were < 18 years old.
  * Aged-matched controls from men attending the Family Planning Association for premarital check-up
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Sperm concentration | up to 3 months
  Sperm concentration

SECONDARY OUTCOMES:
Semen parameters | up to 3 months
  Based on the WHO criteria

OTHER OUTCOMES:
Testicular volume | up to 3 months
  Measured with the Prader orchidometer
Hormonal profile | up to 3 months
  Serum level of testosterone

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, China

IPD SHARING:
Plan to Share IPD: Undecided